CLINICAL TRIAL: NCT00669747
Title: A Phase II Randomized Study Of Intraductal Carboplatin In Women With Ductal Carcinoma In Situ
Brief Title: Study Of Intraductal Carboplatin In Women With Ductal Carcinoma In Situ (DCIS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Windy Hill Medical, Inc. (Industry)
Responsible Party: Windy Hill Medical, Inc. (Ms. Jane Doerr, R.N., Director of Clinical Development), Windy Hill Medical, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCIS-WHM-703M
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Last update posted 2008-10-02 (Estimated); Status verified 2008-10

CONDITIONS: Ductal Carcinoma In Situ
Keywords: Ductal Carcinoma In Situ; DCIS; Breast Cancer; Carboplatin; Intraductal
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms | interventions — Carboplatin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Carboplatin infused into DCIS-involved duct on Days 1 & 15
  Interventions: Drug: Carboplatin i.d. Days 1 & 15
- B (Experimental): Carboplatin infused into DCIS-involved duct Day 1 and Normal Saline infused into DCIS-involved duct on Day 15
  Interventions: Drug: Carboplatin i.d. Day 1; Normal Saline i.d. Day 15
- C (Placebo Comparator): Normal Saline infused into DCIS-involved duct Days 1 & 15
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Carboplatin i.d. Days 1 & 15 — Carboplatin, 10 mg/ml, 10 ml (100 mg) infused into DCIS-involved duct on Days 1 & 15
  Other Names: Paraplatin
  Arms: A
Drug: Carboplatin i.d. Day 1; Normal Saline i.d. Day 15 — Carboplatin 10 mg/ml, 10 ml (100 mg) i.d. DCIS duct on Day 1 Normal Saline, 10 ml i.d. DCIS duct on Day 15
  Other Names: Paraplatin
  Arms: B
Drug: Normal Saline — Normal Saline, 10 ml, i.d. on Days 1 and 15
  Arms: C

SUMMARY:
The primary objective of this study is to compare the safety of 100 mg carboplatin administered intraductally once on Day 1 or twice on Days 1 and 15 in women with ductal carcinoma in situ (DCIS) undergoing surgical management 2 to 4 weeks following the Day 15 intraductal infusion. Secondary objectives are to characterize the biologic and clinical effects with respect to: pharmacokinetics, extent of disease on MRI and mammogram, histopathological assessment of DCIS, and biomarker measurement of Ki-67, TUNEL and G-actin.

DETAILED DESCRIPTION:
This is a randomized, 3-arm, saline-controlled study involving women undergoing surgical management of DCIS. Forty-five (45) women who have been diagnosed with DCIS by core biopsy will receive intraductal administration of either carboplatin or normal saline (NS) into the DCIS-involved breast duct. Thirty (30) patients (i.e., 15 patients per arm) will receive two intraductal infusions of either 100 mg of carboplatin or NS on Days 1 and 15. Fifteen (15) patients will receive an intraductal infusion of 100 mg carboplatin on Day 1 and an intraductal infusion of NS on Day 15. Patients will undergo surgical resection 2 to 4 weeks following the Day 15 intraductal infusion (i.e. 4 to 6 weeks from diagnosis).

The effect of carboplatin on DCIS in the pre-treatment core biopsy specimen and the resection specimen will be assessed. Venous blood samples will be collected for carboplatin PK analysis pre-dose and at 30 minutes, 1, 2, 4, and 8 hours following intraductal infusions on Days 1 and 15.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years of age or older
* Scheduled to undergo surgical resection in 2 weeks or longer
* Pathological diagnosis of DCIS requiring surgical resection
* DCIS diagnosed with core biopsy
* Mammogram within 6 weeks of diagnosis
* Adequate organ function as defined by the following criteria:

Absolute neutrophil count (ANC) ≥ 1500/μl, Platelets ≥ 140,000/μl,Hemoglobin ≥ 12.0 g/dl, Creatinine < 2.0 mg/dl

- Able to sign informed consent

Exclusion Criteria:

* Current diagnosis of invasive or inflammatory breast carcinoma
* DCIS with microinvasion on histology on core needle biopsy
* Palpable mass
* Mass on mammography
* Concurrent anti-cancer therapy
* Prior exposure to carboplatin (related to current or past diagnosis)
* Prior radiation to the breast or chest wall
* Prior areolar or breast surgery which interrupts communication of the ductal systems with the nipple
* Presence of breast implants
* Presence of ulcerating or fungal skin lesions or infection of the breasts
* Pregnant or lactating
* Impaired cardiac function or history of cardiac problems
* Poor nutritional state (as determined by clinician)
* Presence of serious infection
* Scheduled for intraoperative radiation of breast or chest wall
* Allergies to lidocaine or marcaine
* Allergies to imaging dyes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-09 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Compare the safety of 100 mg carboplatin administered intraductally once on Day 1 or twice on Days 1 and 15 in women with ductal carcinoma in situ (DCIS) undergoing surgical management 2 to 4 weeks following the Day 15 intraductal infusion | 2 to 4 weeks following the Day 15 intraductal infusion

SECONDARY OUTCOMES:
characterize i.d. carboplatin pharmacokinetics | 4 -8 weeks
characterize clinical extent of disease on MRI and/or mammogram | 2 - 4 weeks
characterize the histopathological assessment of DCIS | 4 - 10 weeks
Biomarker measurement of Ki-67, TUNEL and G-actin | 4 - 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jane Doerr, RN, MSN, Study Director — Windy Hill Medical, Inc.
Locations (2):
- United States (2):
  - OU Medical Center Laboratory, Oklahoma City, Oklahoma
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Love SM, Barsky SH. Anatomy of the nipple and breast ducts revisited. Cancer. 2004 Nov 1;101(9):1947-57. doi: 10.1002/cncr.20559. PMID 15382093
- [Background] Li CI, Daling JR, Malone KE. Age-specific incidence rates of in situ breast carcinomas by histologic type, 1980 to 2001. Cancer Epidemiol Biomarkers Prev. 2005 Apr;14(4):1008-11. doi: 10.1158/1055-9965.EPI-04-0849. PMID 15824180
- [Background] Khan SA, Wiley EL, Rodriguez N, Baird C, Ramakrishnan R, Nayar R, Bryk M, Bethke KB, Staradub VL, Wolfman J, Rademaker A, Ljung BM, Morrow M. Ductal lavage findings in women with known breast cancer undergoing mastectomy. J Natl Cancer Inst. 2004 Oct 20;96(20):1510-7. doi: 10.1093/jnci/djh283. PMID 15494601